CLINICAL TRIAL: NCT07356089
Title: Twiist Postmarket Surveillance Study in Adults and Youth With Type 1 Diabetes
Brief Title: Twiist Postmarket Surveillance Study for Type 1 Diabetes
Acronym: twiist-PS
Status: Recruiting | Type: Observational
Sponsor: Deka Research and Development (Industry)
Collaborators: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Other Study IDs: DKPI-00741-001
Record Dates: First submitted 2026-01-06; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes (T1D); Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Pediatric Postmarket Surveillance: Yes | US Export: No

GROUPS / COHORTS (1):
- twiist users
  Interventions: Device: twiist Automated Insulin Delivery System

INTERVENTIONS:
Device: twiist Automated Insulin Delivery System — twiist(TM) system includes a novel insulin pump, a CGM sensor, and the glycemic-control algorithm

SUMMARY:
The goal of this surveillance study is to collect real-world data on adults and youth with type 1 diabetes (T1D) using twiist(TM) for insulin delivery.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent (or a parent or other legally authorized representative)
* Age ≥ 6 years old
* Diagnosis of T1D
* Currently using twiist AID system, with initiation of twiist within 90 days of enrollment
* Willing to only use an insulin approved for the pump
* Residing in United States
* Willing to use twiist in accordance with the user manual
* Willing to have the study use the twiist data and any information that has been provided to Sequel Medtech, LLC or customer support since twiist was started
* Willing to complete surveys at the beginning of the study and then monthly for 12 months
* Willing to be contacted if clarification or further information is needed for any events reported on a survey or to customer support
* Willing to provide medical records or sign a record release for any hospitalizations
* Has cell service or if not, will have access to WIFI at least once a week
* For females, not pregnant or planning pregnancy in the next 12 months
* Able to speak and read English
* Able to obtain documentation of HbA1c result obtained within 6 months prior to twiist initiation

Exclusion Criteria:

* Any form of diabetes other than T1D
* Receiving dialysis for end-stage renal disease

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who are diagnosed with Type 1 Diabetes, are at least 6 years old, and have been prescribed and are currently using the twiist system.
Sampling Method: Non-Probability Sample
Enrollment: 1875 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Severe hypoglycemia events | From enrollment to the end of participation at 12 months
  Severe hypoglycemia events with cognitive impairment sufficient to require the assistance of a third party for treatment

SECONDARY OUTCOMES:
Severe hypoglycemia events associated with seizure or loss of consciousness | From enrollment to the end of participation at 12 months
Diabetic ketoacidosis | From enrollment to the end of participation at 12 months
Hospitalizations related to use of twiist | From enrollment to the end of participation at 12 months
Unanticipated adverse device effects | From enrollment to the end of participation at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jaeb Center for Health Research, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No